CLINICAL TRIAL: NCT00858299
Title: The Change of Urinary Angiotensinogen Excretion After Valsartan Treatment in Chronic Kidney Diseases Patients With Persistent Proteinuria
Brief Title: The Change of Urinary Angiotensinogen Excretion After Valsartan Treatment in Patients With Persistent Proteinuria
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Yoon-Goo Kim, Division of Nephrology, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2008-07-089
Record Dates: First submitted 2009-03-05; First posted 2009-03-09 (Estimated); Last update posted 2009-03-09 (Estimated); Status verified 2009-03

CONDITIONS: Chronic Kidney Disease; Proteinuria
Keywords: proteinuria; chronic kidney disease; renin-angiotensin system; angiotensinogen
MeSH Terms: conditions — Renal Insufficiency, Chronic; Proteinuria | interventions — Valsartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- valsartan (Experimental)
  Interventions: Drug: valsartan

INTERVENTIONS:
Drug: valsartan — 160 mg oral once in a day for initial 8 weeks and 320 mg, oral, once in a day for subsequent 16 weeks

SUMMARY:
This study is a multicenter, prospective, interventional study. It does not have a control group. All participants will receive 160 mg valsartan for 8 weeks. Among them, the patients with persistent proteinuria (defined as proteinuria more than 1 g/g after 8 weeks treatment of valsartan) will receive 320 mg valsartan for further 16 weeks. Participants who did not receive any ACEI or ARB previously will have a titration period for 4 weeks (80 mg for 4 weeks, 160 mg for 4 weeks, and then 320 mg for 16 weeks).

The investigators will evaluate the change of urinary angiotensinogen excretion between at baseline, at 8 weeks, and 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Chronic kidney disease patients with

  * proteinuria of 1 - 10 g/day,
  * stable and controlled blood pressure (100/60 mmHg - 160/100 mmHg),
  * stable renal function with GFR ≥ 30 mL/min/ m2,
  * diabetes or non-diabetes

Exclusion Criteria:

* Uncontrolled diabetes (defined as HbA1c > 9.0%)
* Immunosuppressive treatment within 6 months
* Intractable edema
* Hyperkalemia (>5.5 mEq/L) or Hypokalemia (< 3.5 mEq/L)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2009-03; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
The percent change of urinary angiotensinogen excretion between at baseline and at 24 weeks after valsartan treatment. | 4 weeks of screening periods + 24 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Yoon-Goo Kim, Professor, Principal Investigator — Division of Nephrology, Samsung Medical Center
Locations (1):
- Division of Nephrology, Samsung Medical Center, Seoul, Seoul, South Korea